CLINICAL TRIAL: NCT01961401
Title: Acute Effects of Moderate Versus High Intensity Exercise on Insulin Sensitivity in Pregnant Women With and Without Gestational Diabetes Mellitus
Brief Title: Acute Effects of Moderate Versus High Intensity Exercise on Insulin Sensitivity in Gestational Diabetes Mellitus
Acronym: GDMakutt
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to recruitment problems
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012/1021
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Diabetes, Gestational
Keywords: exercise; exercise therapy; insulin resistance
MeSH Terms: conditions — Diabetes, Gestational; Motor Activity; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High intensity exercise (Experimental): High intensity, short duration exercise on bike
  Interventions: Behavioral: exercise
- Moderate exercise (Experimental): Moderate intensity exercise training on bike
  Interventions: Behavioral: exercise
- No exercise (No Intervention): No exercise, resting in the lab

INTERVENTIONS:
Behavioral: exercise
  Arms: High intensity exercise; Moderate exercise

SUMMARY:
Exercise training is recognized as effective in preventing and treating many chronic metabolic disorders (1), and long-term exercise programmes have similar effects on glucose control as long-term drug or insulin therapy in type 2 diabetic patients (2). The precise intensity and volume of aerobic exercise needed to produce the most wanted effects on targeted risk factors for subjects at risk of/with established type 2 diabetes, is still uncertain. In this study the investigators will investigate the acute effects of a single bout of moderate versus high intensity exercise on insulin sensitivity in pregnant women with and without gestational diabetes mellitus (GDM). The investigators think that very short bouts of high intensity exercise can be a way to reduce blood glucose in these women.

ELIGIBILITY:
Inclusion Criteria:

* pregnant
* Gestational diabetes mellitus or normal glucose tolerance
* able to exercise

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2013-01; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | 1 day
  insulin sensitivity index, as described by Matsuda and DeFronzo. This calculation uses the fasting plasma glucose and plasma insulin, and the average plasma glucose and insulin values over the 30, 60, 90, and 120 minutes after an oral glucose tolerance test (OGTT), and is calculated as:. 10 000/√[fasting glucose x fasting insulin) x (mean glucose during OGTT x mean insulin during OGTT)]. We will use a carbohydrate rich meal instead of a classic oral glucose tolerance test with glucose in water.

CONTACTS AND LOCATIONS:
Overall Officials: trine Moholdt, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of circulation and medical imaging, Trondheim, Norway